CLINICAL TRIAL: NCT00013663
Title: A Randomized Controlled Study Testing the Efficacy of Immunotherapies to Control Plasma HIV RNA Concentrations Upon Interruption of Highly Active Antiretroviral Therapy
Brief Title: Immune Therapies and Anti-HIV Therapy Withdrawal in Controlling Viral Load
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: New York Presbyterian Hospital (Other)
Masking: Double | Purpose: Treatment
Other Study IDs: B012; 0900-397; NCT00034099 (obsolete NCT alias)
Record Dates: First submitted 2001-03-27; First posted 2001-08-31 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2006-06

CONDITIONS: HIV Infections
Keywords: Virus Replication; HIV-1; AIDS Vaccines; RNA, Viral; Avipoxvirus; Genetic Vectors; Viral Load; aldesleukin; Antiretroviral Therapy, Highly Active; HIV Therapeutic Vaccine; Treatment Interruption
MeSH Terms: conditions — HIV Infections | interventions — aldesleukin

INTERVENTIONS:
Biological: ALVAC(2)120(B,MN)GNP (vCP1452)
Drug: Aldesleukin

SUMMARY:
The purpose of this study is to determine if HIV-specific canarypox vaccine and/or interleukin-2 (IL-2) will control viral load (amount of HIV in the blood) after HIV treatment is withdrawn for a certain time period.

DETAILED DESCRIPTION:
Step I: In addition to continuing HAART, patients are randomized into 1 of the following 4 arms:

A: Immunization placebo; B: Immunization with the canarypox HIV-vaccine (vCP1452); C: Daily low-dose IL-2 + immunization placebo; or D: Daily low-dose IL-2 + canarypox HIV-vaccine (vCP1452). Patients on Arms A, B, C, and D receive vaccine (or vaccine placebo) injections at Weeks 0, 4, 8, and 12. Patients on Arms C and D receive IL-2 by self-injection. HAART is not provided as part of this study.

Step II: Patients on all arms (A, B, C, and D) who meet inclusion criteria advance to Step II and interrupt HAART for a minimum of 12 weeks. The efficacy of these immunological therapies will be determined by monitoring the dynamics of viral rebound upon cessation of antiviral therapy. After 12 weeks of Step II, patients whose viral load remains below 30,000 copies/ml remain on Step II, off HAART, and continue weekly viral load monitoring. Patients will not terminate Step II or resume HAART unless and until their viral load increases to more than 30,000 copies/ml on 3 successive determinations, or their CD4 count decreases to less than 200 cells/mm3 or less than 50 percent of the baseline CD4+ T cell concentration on 2 successive occasions.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are more than 18 years old.
* Have been receiving their current HAART (2 or more anti-HIV drugs in combination) for more than 6 consecutive months.
* Have a CD4 count of 200 cells/microL or more within the 12 months prior to entering the study and 400 cells/microL or more on 2 occasions at least 2 weeks apart within 30 days of entry.
* Have never had a viral load higher than 2 million molecules/ml and have had the viral load controlled with HAART to less than 50 molecules/ml on 2 occasions at least 2 weeks apart within 30 days of entry.
* Have not had virologic failure on the current HAART regimen.
* Have a negative urine pregnancy test within 14 days of entering the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a current AIDS-defining illness.
* Have had failure of the current HAART regimen (viral load higher than 10,000 molecules/ml).
* Have a history of using agents affecting the immune system.
* Have active uncontrolled heart disease.
* Have had IL-2 therapy within 4 weeks of entering the study.
* Have received other treatment that affects the immune system within 4 weeks of entry.
* Have a history of a cancer requiring chemotherapy.
* Have untreated thyroid disease, within 4 weeks of entering the study.
* Have uncontrolled allergic disorders or autoimmune diseases, including asthma, inflammatory bowel disease, and psoriasis.
* Abuse substances that may interfere with the ability to follow study requirements.
* Are allergic to eggs.
* Have hepatitis B or hepatitis C.
* Are pregnant or breast-feeding.
* Work in close contact with canaries, such as a job at breeding farms or bird shops.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92
Dates: Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Mean log10 viral load for each experimental group from the average of 5 values obtained during Weeks 21 to 25 (8 to 12 weeks following HAART interruption

SECONDARY OUTCOMES:
Proportion of participants who relapse during the first 12 weeks following stopping of HAART
length of time to the termination of Step II among participants
changes in frequency, activation state, and HIV-specific functional capacity of T and NK cells in blood, as monitored by expression of intracellular cytokines during the first 12 weeks after stopping HAART, with respect to termination of Step II

CONTACTS AND LOCATIONS:
Overall Officials: Kendall A. Smith, MD, Principal Investigator — Division of Immunology, Department of Medicine, Weill Medical College, Cornell University
Locations (1):
- New York Hosp - Cornell Med Ctr, New York, New York, United States